CLINICAL TRIAL: NCT01103596
Title: Evaluation of the Public Health Interest of Kaletra: Impact on Resistance to ARVs - EOLE
Brief Title: Evaluation of the Public Health Interest of Kaletra: Impact on Resistance to Antiretrovirals (ARVs)
Acronym: EOLE
Status: Completed | Type: Observational
Sponsor: Abbott (Industry)
Collaborators: Readitwell (Unknown); Lincoln Medical and Mental Health Center (Other)
Responsible Party: Sponsor
Other Study IDs: P06-124
Record Dates: First submitted 2010-02-24; First posted 2010-04-14 (Estimated); Last update posted 2011-12-14 (Estimated); Status verified 2011-12

CONDITIONS: HIV Infection
Keywords: Evaluation of the impact of Kaletra on antiretroviral resistance
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — Frozen plasma for determination of Lopinavir/ritonavir (LPV/r) Cmin
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- HIV-infected patients, 1st wave: HIV-infected ARV-experienced patients treated by a combination including Kaletra
- HIV-infected patients, 2nd wave: HIV-infected ARV-experienced patients treated by a combination including Kaletra

SUMMARY:
The purpose of this study is to evaluate, in patients in at least the second protease inhibitor (PI) line, the virological failures under Kaletra® and their consequences on protease and reverse transcriptase genotypes

DETAILED DESCRIPTION:
The purpose of this study is to evaluate, in patients in at least the second PI line, the virological failures under Kaletra® and their consequences on protease and reverse transcriptase genotypes:

* Characterisation of the changes in the resistance genotype in protease and reverse transcriptase,
* Description of the nature and frequency of selected mutations under Kaletra®,
* Description of the predictive factors for mutations and of the impact they could have on other PIs used as maintenance treatment (analysis based on available algorithms).

EOLE is a prospective, multicentre observation study offered to French virology laboratories and involving clinical teams .

It is a transversal study with retrospective data collection for patients meeting the study criteria (virological failure under Kaletra® after at least first line PI treatment).

The study comprises two enrolment periods, separated by an interval of one year, over a period ranging from 2007 to 2011. During this period, virological failures under Kaletra® are identified. For each period, the virologists collect data only from the moment when virological failure under Kaletra® is identified.

The first wave of data collection is now completed and occurred from December 5, 2007 to July 03, 2009.

It is not planned to collect follow-up data in connection with alternative treatment with other antiretrovirals after failure under Kaletra®.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged under 18 years,
* Pre-treated by at least one protease inhibitor (PI) line,
* In therapeutic failure of the antiretroviral (ARV) maintenance treatment containing Kaletra®.

Therapeutic failure is defined by a viral load> 50 copies/ml after at least three months' treatment with an ARV combination containing Kaletra®, always provided that genotyping is possible .

Exclusion Criteria:

* Patients having received less than three months of Kaletra®,
* Patients for whom the genotype information before starting Kaletra® and at the time of the failure of Kaletra® was not available,
* Patients receiving another protease inhibitor (PI) concomitantly with Kaletra®.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Virology laboratories
Sampling Method: Non-Probability Sample
Enrollment: 94 (Actual)
Dates: Start 2008-03; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
Genotype for resistance determination | Over the duration of the enrollment for each wave, over a total period of 18 months
Description of the predictive factors for mutations and of the impact they could have on other protease inhibitors (PIs) used as maintenance treatment (analysis based on available algorithms). | Over the duration of the enrollment for each wave, over a total period of 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Isabelle Cohen Codar, PharmD, Study Director — Abbott France
Locations (19):
- France (19):
  - Site Reference ID/Investigator# 27801, Angers
  - Site Reference ID/Investigator# 27799, Bordeaux
  - Site Reference ID/Investigator# 27790, Grenoble
  - Site Reference ID/Investigator# 27796, Lille
  - Site Reference ID/Investigator# 27786, Montpellier
  - Site Reference ID/Investigator# 27800, Nantes
  - Site Reference ID/Investigator# 27798, Nice
  - Site Reference ID/Investigator# 27792, Nîmes
  - Site Reference ID/Investigator# 5595, Paris
  - Site Reference ID/Investigator# 27787, Paris
  - Site Reference ID/Investigator# 27797, Paris
  - Site Reference ID/Investigator# 27783, Paris
  - Site Reference ID/Investigator# 27802, Paris
  - Site Reference ID/Investigator# 27785, Paris
  - Site Reference ID/Investigator# 27791, Rennes
  - Site Reference ID/Investigator# 27788, Rouen
  - Site Reference ID/Investigator# 27789, Toulon
  - Site Reference ID/Investigator# 27794, Toulouse
  - Site Reference ID/Investigator# 27784, Villejuif